CLINICAL TRIAL: NCT00614211
Title: A Phase III Randomized Clinical Trial of Laparoscopic or Robotic Radical Hysterectomy Versus Abdominal Radical Hysterectomy in Patients With Early Stage Cervical Cancer
Brief Title: Laparoscopic Approach to Cervical Cancer
Acronym: LACC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queensland Centre for Gynaecological Cancer (Other Government)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LACC001
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Cervical Cancer
Keywords: Cervix; Cervical; Cancer; Carcinoma; Radical hysterectomy; Hysterectomy; Laparoscopy; Laparoscopic; Robotic; Squamous Cell; Adenosquamous; Adenocarcinoma; Lymphatic Mapping; IOLM; SPECT; Sentinel Node; Uterine cervix
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasms; Carcinoma; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Total Abdominal Radical Hysterectomy
  Interventions: Procedure: Total Abdominal Radical Hysterectomy
- 2 (Experimental): Total Laparoscopic or Robotic Radical Hysterectomy
  Interventions: Procedure: Total Laparoscopic or Robotic Radical Hysterectomy

INTERVENTIONS:
Procedure: Total Abdominal Radical Hysterectomy — In a radical hysterectomy the uterus, the upper one to two centimetres of the vagina and the soft tissues around the cervix are excised.
  Other Names: TARH; Open radical hysterectomy
  Arms: 1
Procedure: Total Laparoscopic or Robotic Radical Hysterectomy — In a radical hysterectomy the uterus, the upper one to two centimetres of the vagina and the soft tissues around the cervix are excised.
  Other Names: TLRH; TRRH; Keyhole radical hysterectomy
  Arms: 2

SUMMARY:
The goal of this clinical research study is to compare the long-term outcomes of different surgical methods for the treatment of cervical cancer. The long-term outcome of a total abdominal radical hysterectomy (TARH) will be compared against laparoscopy. In this study, the laparoscopy will be done with or without robotic technology.

DETAILED DESCRIPTION:
Primary Objective:

To compare disease-free survival amongst patients who undergo a total laparoscopic (TLRH) or robotic radical hysterectomy (TRRH) verses those who undergo a total abdominal radical hysterectomy (TARH) for early stage cervical cancer.

Secondary Objectives:

* Compare patterns of recurrence between arms.
* Compare treatment-associated morbidity within 6 months from surgery.
* Compare the cost effectiveness of TLRH/TRRH versus TARH
* Compare the impact on Quality of Life (QOL) between arms.
* Assess pelvic floor function
* Compare overall survival between arms
* Determine the feasibility of sentinel lymph node biopsy in this group of patients

RATIONALE FOR STUDY DESIGN Total abdominal radical hysterectomy (TARH) and pelvic lymph node dissection (± aortic lymph node dissection ± postoperative [chemo-] radiotherapy) is the current standard treatment for early cervical cancer. While this is an accepted effective treatment, a laparotomy is highly invasive, visibly scarring and is associated with tissue trauma, blood loss and a significant risk of wound and infectious adverse events . Additionally, radical hysterectomy by laparotomy is associated with an average hospital stay of approximately 5 to 7 days and an average recovery period (from surgery) of 5 to 6 weeks.

Laparoscopic techniques have been demonstrated to be feasible and safe with previous retrospective studies on TLH showing encouraging results . In a number of retrospective and prospective, non-controlled series the incidence of treatment-related morbidity was less in patients who had a laparoscopic hysterectomy compared to patients who underwent a TAH . Retrospective data suggest that the recurrence rate and patterns of recurrence are similar in patients who had a laparoscopic or an open approach .

Treatment recommendations ideally are based on prospective, randomized trials comparing the current standard technique (TARH) with the proposed better technique (TLRH). However, there are currently no prospective studies available which directly compare TLRH against the standard treatment of TARH in regards to disease-free or overall survival.

The proposed clinical trial will be biphasic. The primary outcome variable in stage 1 will be feasibility of recruitment as determined by overall trial recruitment. Following completion of Stage 1, the data of this study will become the basis for assessing recurrence and disease-free survival in the Stage 2 design.

RATIONALE FOR THE QUALITY OF LIFE Retrospective studies suggest equivalency between the laparoscopic and open approaches to radical hysterectomy in regards to surgical specimens obtained and likely disease-free and overall survivals . Thus, quality of life could be seen as one of the most significant factors in recommending one approach over the other and therefore an extremely important endpoint for this protocol. In the GOG LAP-2 protocol , a trial evaluating a comparison between hysterectomy by laparotomy or laparoscopy, the investigators found equivalency adequacy of the two surgical approaches however a significant difference in short term quality of life favoring laparoscopy. As expected, patients who underwent laparoscopy had a faster return to baseline functioning compared with those patients who had undergone laparotomy which translated into improved short-term quality of life. By 6 months, however, patients in both cohorts were reporting equivalent quality of life parameters. Quality of life surveys employed with this Phase III clinical trial will encompass important endpoints such as postoperative pain and related symptoms using the MD Anderson Symptom Assessment Index (MDSAI), as well as cancer specific Functional Assessment of Cancer Therapy (FACT-Cx) and the general 12-Item Short-Form Health Survey (SF-12).

RATIONALE FOR LYMPHATIC MAPPING Published experience with the techniques for lymphatic mapping and sentinel lymph node detection in women with cervical cancer has been very limited. To date, no single study has enrolled more than 100 patients undergoing lymphatic mapping as part of their surgical treatment for cervical cancer. In fact, the majority of studies report on less than 50 patients. In addition, this procedure has not yet been shown to be viable in a multi-institutional setting. The limitations of previously published reports are important as these techniques are associated with a significantly high learning curve with early procedures less successful than later ones. This study will provide us the opportunity to enroll large numbers of patients for validation of intraoperative lymphatic mapping in women with cervical cancer in an international, multi-institutional setting.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary adenocarcinoma, squamous cell carcinoma or adenosquamous carcinoma of the uterine cervix;
* Patients with Histologically confirmed stage IA1 (with lymph vascular invasion), stage IA2, or stage IB1 disease
* Patients undergoing either a Type II or III radical hysterectomy (Piver Classification)
* Patients with adequate bone marrow, renal and hepatic function:
* ECOG Performance Status of 0 or 1.
* Patient must be suitable candidates for surgery.
* Patients who have signed an approved Informed Consent
* Patients with a prior malignancy allowed if > 5 years ago with no current evidence of disease
* Females, aged 18 years or older
* Negative serum pregnancy test within <30 days of surgery in pre-menopausal women and women < 2 years after the onset of menopause

Exclusion Criteria:

* Any histology other than adenocarcinoma, squamous cell carcinoma or adenosquamous carcinoma of the uterine cervix;
* Tumor size greater than 4 cm;
* FIGO stage II-IV;
* Patients with a history of pelvic or abdominal radiotherapy;
* Patients who are pregnant;
* Patients with contraindications to surgery;
* Patients with evidence of metastatic disease by conventional imaging studies, enlarged pelvic or aortic lymph nodes > 2cm; or histologically positive lymph nodes
* Unfit for Surgery: serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator);
* Patients unable to withstand prolonged lithotomy and steep Trendelenburg position
* Patient compliance and geographic proximity that do not allow adequate follow-up

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 636 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2022-03 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Disease free survival | 5 years from surgery
  Compare treatment equivalence

SECONDARY OUTCOMES:
Patterns of recurrence | 5 years from surgery
  date and localization of 1st recurrence as confirmed histologically - Compare patterns between groups
Costs | 6 months from surgery
  Compare costs between groups
Quality of life Questionnaires | 6 months from surgery
  Compare QoL between groups
Pelvic Floor Distress Inventory Questionnaire | 5 years from surgery
  Compare PFDI between groups
Overall survival | 5 years from surgery
  Compare between groups
Feasibility of sentinel lymph node biopsy | Intra-operatively
  Compare between groups
Intra-operative, peri-operative, post-operative and long term treatment related morbidity | 6 months from surgery
  Compare these between groups

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Ramirez, M.D., Study Chair — M.D. Anderson Cancer Center; Andreas Obermair, MD, Study Chair — Queensland Centre for Gynecological Cancer; Michael Frumovitz, M.D., Study Chair — M.D. Anderson Cancer Center
Locations (33):
- United States (6):
  - Greater Baltimore Medical Centre, Baltimore, Maryland
  - Women's Cancer Centre Nevada, Las Vegas, Nevada
  - St Luke's - Roosevelt Hospital Center, New York, New York
  - Peggy and Charles Stephenson Oklahoma Cancer Center, Oklahoma City, Oklahoma
  - M.D. Anderson Cancer Center, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin
- Misericordia Hospital, Córdoba, Argentina
- Australia (6):
  - The Wesley Hospital, Auchenflower, Queensland
  - Greenslopes Private Hospital, Greenslopes, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Mater Health Services, South Brisbane, Queensland
  - The Townsville Hospital, Townsville, Queensland
  - Saint John of God, Subiaco, Western Australia
- Brazil (4):
  - Erastus Gaertner Hospital, Curitiba, Paraná
  - Barretos Cancer Hospital, Barretos, São Paulo
  - Instituto Brasileiro de Controlle do Cancer, Brás, São Paulo
  - Albert Einstein Hospital, Morumbi, São Paulo
- University Hospital Pleven Center of Oncology Gynaecology, Pleven, Bulgaria
- Princess Margaret Hospital, Toronto, Ontario, Canada
- China (3):
  - The First Affilated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Affliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang
- Institito De Cancerologia Clinica Las Americas, Antioquia, Medellin, Colombia
- Italy (4):
  - Alessandro Manzoni Hospital, Lecco, Milan
  - San Gerardo Hospital, Monza, Milan
  - Catholic University of the Sacred Heart, Milan, Rome
  - European Institute of Oncology, Milan
- Instituto Nacional de Cencerologia, Tlalpan, Mexico City, Mexico
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Surquillo, Peru
- Gyneco-Oncologico Hospital HIMA, Caguas, San Pablo, Puerto Rico
- South Korea (3):
  - Korea Cancer Hospital, Goyang-si, Seoul
  - Seoul National University - Department of Obstetrics and Gynecology, Ihwa-dong, Seoul
  - ASAN Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Obermair A, Gebski V, Frumovitz M, Soliman PT, Schmeler KM, Levenback C, Ramirez PT. A phase III randomized clinical trial comparing laparoscopic or robotic radical hysterectomy with abdominal radical hysterectomy in patients with early stage cervical cancer. J Minim Invasive Gynecol. 2008 Sep-Oct;15(5):584-8. doi: 10.1016/j.jmig.2008.06.013. PMID 18722970
- [Derived] Ramirez PT, Robledo KP, Frumovitz M, Pareja R, Ribeiro R, Lopez A, Yan X, Isla D, Moretti R, Bernardini MQ, Gebski V, Asher R, Behan V, Coleman RL, Obermair A. LACC Trial: Final Analysis on Overall Survival Comparing Open Versus Minimally Invasive Radical Hysterectomy for Early-Stage Cervical Cancer. J Clin Oncol. 2024 Aug 10;42(23):2741-2746. doi: 10.1200/JCO.23.02335. Epub 2024 May 29. PMID 38810208
- [Derived] Tanaka T, Ueda S, Miyamoto S, Hashida S, Terada S, Konishi H, Kogata Y, Taniguchi K, Komura K, Ohmichi M. Comparison of Prognosis between Minimally Invasive and Abdominal Radical Hysterectomy for Patients with Early-Stage Cervical Cancer. Curr Oncol. 2022 Mar 24;29(4):2272-2283. doi: 10.3390/curroncol29040185. PMID 35448159
- [Derived] Frumovitz M, Obermair A, Coleman RL, Pareja R, Lopez A, Ribero R, Isla D, Rendon G, Bernardini MQ, Buda A, Moretti-Marquez R, Zevallos A, Vieira MA, Zhu T, Land RP, Nicklin J, Asher R, Robledo KP, Gebski V, Ramirez PT. Quality of life in patients with cervical cancer after open versus minimally invasive radical hysterectomy (LACC): a secondary outcome of a multicentre, randomised, open-label, phase 3, non-inferiority trial. Lancet Oncol. 2020 Jun;21(6):851-860. doi: 10.1016/S1470-2045(20)30081-4. PMID 32502445
- [Derived] Ramirez PT, Frumovitz M, Pareja R, Lopez A, Vieira M, Ribeiro R, Buda A, Yan X, Shuzhong Y, Chetty N, Isla D, Tamura M, Zhu T, Robledo KP, Gebski V, Asher R, Behan V, Nicklin JL, Coleman RL, Obermair A. Minimally Invasive versus Abdominal Radical Hysterectomy for Cervical Cancer. N Engl J Med. 2018 Nov 15;379(20):1895-1904. doi: 10.1056/NEJMoa1806395. Epub 2018 Oct 31. PMID 30380365
- See also: QCGC Research — http://www.gyncan.org/
- See also: Cancer Treatment and Research Centre — http://www.mdanderson.org